CLINICAL TRIAL: NCT00326456
Title: Phase III Randomized Multicentre Trial of Carboplatin + Liposomal Doxorubicin vs Carboplatin + Paclitaxel in Patients With Ovarian Cancer
Brief Title: MITO-2: A Study Comparing 2 Chemotherapy Regimens (Carboplatin/Liposomal Doxorubicin vs Carboplatin/Paclitaxel) in Patients With Ovarian Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MITO-2; 2005-004453-98 (EudraCT Number)
Record Dates: First submitted 2006-05-15; First posted 2006-05-16 (Estimated); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; chemotherapy; first-line
MeSH Terms: conditions — Ovarian Neoplasms | interventions — liposomal doxorubicin; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- carboplatin and liposomal doxorubicin (Experimental)
  Interventions: Drug: liposomal doxorubicin; Drug: carboplatin
- carboplatin and paclitaxel (Active Comparator)
  Interventions: Drug: carboplatin; Drug: paclitaxel

INTERVENTIONS:
Drug: liposomal doxorubicin — 30 mg/m2 gieven intravenously on day 1 every 3 weeks
  Arms: carboplatin and liposomal doxorubicin
Drug: carboplatin — AUC 5 intravenously on day 1 every 3 weeks
Drug: paclitaxel — 175 mg/m2 intravenously on day 1 every 3 weeks
  Arms: carboplatin and paclitaxel

SUMMARY:
The purpose of this study is to compare the effectiveness (progression free survival) of the experimental combination of carboplatin + liposomal doxorubicin with the standard combination of carboplatin + paclitaxel in first line treatment of patients with ovarian cancer.

Secondary objectives are to evaluate overall survival, quality of life, objective response rate, and toxicity.

DETAILED DESCRIPTION:
Ovarian cancer is the second most frequent and the most deadly gynaecologic cancer. The high mortality rate is due to the late diagnosis of this malignancy that often develops without symptoms, as well as to limited results in treatment of the disease. Patients may respond well initially to chemotherapy, but the vast majority of patients will experience a progression of the disease. The poor long term results in the standard treatment available today for first-line chemotherapy of ovarian cancer make research into new, more beneficial treatment strategies necessary. The proven efficacy of liposomal doxorubicin in second line treatment, where it is the first drug to have shown some significant benefit in terms of survival, and the possibility of easily combining it with full doses and normal use of carboplatin, encourages the testing of the effectiveness of the combination of carboplatin and liposomal doxorubicin in first line treatment.

Patients enrolled into this study will be randomly assigned to one of two treatment groups:

· Standard therapy consisting of 6 cycles of chemotherapy:

* carboplatin AUC 5 given intravenously on day 1 every 3 weeks AND
* paclitaxel 175 mg/m2 given intravenously on day 1 every 3 weeks

OR

· Experimental therapy consisting of 6 cycles of chemotherapy:

* carboplatin AUC 5 given intravenously on day 1 every 3 weeks AND
* liposomal doxorubicin 30 mg/m2 given intravenously on day 1 every 3 weeks

ELIGIBILITY:
Inclusion Criteria:

* Cytologic / histologic diagnosis of stage Ic-IV ovarian cancer
* Indication for chemotherapy treatment
* Age 75 years or less
* Life expectancy of at least 3 months

Exclusion Criteria:

* Previous or concomitant malignant neoplasia (not including basocellular or spinocellular skin carcinoma or in-situ carcinoma of the uterine cervix, provided they are being adequately treated)
* Performance status (ECOG) > 2
* Previous chemotherapy treatment
* Heart disease (heart failure, myocardial heart attack within 6 months prior to randomization, atrioventricular block of any degree, serious arrhythmia)
* Leukocytes < 4000/mm3, neutrophils < 2000/mm3, platelets < 100000/mm3
* Impaired renal function (creatinine > 1.25 times the upper normal limit) or liver function (SGOT or SGPT > 1.25 times the upper normal limit)
* Present or suspected hemorrhagic syndromes
* Uncooperative and/or unreliable patients
* Patient's inability to access the center
* Refusal of informed consent

Max Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 820 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | at 2 years

SECONDARY OUTCOMES:
overall survival | 4 years
quality of life | at baseline and every 3 weeks during treatment
objective response rate | at 9 and 18 weeks after starting study therapy
adverse events | every 3 weeks during chemotherapy
  according to CTCAE criteria

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Pignata, M.D., Ph.D, Principal Investigator — National Cancer Institute, Naples; Francesco Perrone, M.D., Ph.D, Principal Investigator — National Cancer Institute, Naples
Locations (38):
- Italy (36):
  - Clinica Malzoni, Reparto di Ginecologia Oncologica, Avellino, AV
  - Azienda Ospedaliera S. Giuseppe Moscati, U.O. di Oncologia Medica, Monteforte Irpino, AV
  - Ospedale Regionale Miulli, Divisione Medicina Interna Sezione Oncologica, Acquaviva delle Fonti, BA
  - IRCCS Oncologico Bari, Oncologia Medica, Bari, BA
  - Istituto Oncologico di Bari, U.O. di Oncologia Medica e Sperimentale, Bari, BA
  - Ospedale Riuniti di Bergamo, U.O. di Ostetricia e Ginecologia, Bergamo, BG
  - Ospedale Fatebenefratelli, U.O. di Oncologia, Benevento, BN
  - Ospedale di Bentivoglio, Bentivoglio, BO
  - Ospedale Bellari, U.O. di Oncologia, Bologna, BO
  - Ospedale di Budrio, Budrio, BO
  - Policlinico Universitario, Oncologia Medica II, Cagliari, CA
  - Università Cattolica del Sacro Cuore, Dipartimento di Oncologia, Campobasso, CB
  - Ospedale Mariano Santo, U.O. di Oncologia Medica, Cosenza, CS
  - Ospedale Cannizzaro, Divisione di Ostetricia e Ginecologia, Catania, CT
  - Azienda Ospedaliera Universitaria Acrispedale Sant'Anna, Ferrara, FE
  - Ospedale Pierantoni, Divisione di Oncologia Medica, Forlì, FO
  - Azienda Ospedaliera Carlo Poma, Divisione di Oncologia ed Ematologia, Mantova, MN
  - Ospedale Ramazzini, Day Hospital Oncologico, Carpi, MO
  - Policlinico Universitario P. Giaccone, Palermo, PA
  - Ospedale M. Ascoli, Palermo, PA
  - Casa di Cura La Maddalena S.p.A., Dipartimento Oncologico, Palermo, PA
  - Ospedale S. Massimo, Day Hospital Oncologico, Penne, PE
  - Centro di Riferimento Oncologico, Divisione di Oncolgia Medica C, Aviano, PN
  - Azienda Ospedaliera S. Maria degli Angeli, Servizio di Oncologia, Pordenone, PN
  - Ospedale Civile di Faenza, Divisione di Oncologia Medica, Faenza, RA
  - Azienda Ospedaliera Bianchi Melacrino Morelli Ospedale Riuniti, Divisione di Oncologia Medica, Reggio Calabria, RE
  - Ospedale degli Infermi, U.O. Oncologia Medica, Rimini, RI
  - Ospedale Civile Umberto I, Day Hospital Oncoematologico, Nocera Inferiore, SA
  - Ospedale S. Chiara, U.O. di Oncologia Medica, Trento, TN
  - Ospedale S. Anna, Day Hospital Oncologico Divisione A, Torino, TO
  - Ospedale S. Bortolo ULSS 6, U.O. di Oncologia Medica, Vicenza, VI
  - Azienda Ospedaliera D. Cotugno, Napoli
  - Istituto Nazionale dei Tumori , Divisione di Oncologia Medica B, Napoli
  - Istituto Nazionale dei Tumori, Divisione di Oncologia Medica C, Napoli
  - Istituto Regina Elena, Divisione di Oncologia Medica, Roma
  - Ospedale S. Giovanni Calibita Gatebenefratelli, Roma
- CHC Maternidade Bissaya-Barreto, Gynecology Unit, Coimbra, Portugal
- Istanbul University Medical Oncology, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Pignata S, Scambia G, Savarese A, Breda E, Scollo P, De Vivo R, Rossi E, Gebbia V, Natale D, Del Gaizo F, Naglieri E, Ferro A, Musso P, D'Arco AM, Sorio R, Pisano C, Di Maio M, Signoriello G, Annunziata A, Perrone F; MITO Investigators. Safety of a 3-weekly schedule of carboplatin plus pegylated liposomal doxorubicin as first line chemotherapy in patients with ovarian cancer: preliminary results of the MITO-2 randomized trial. BMC Cancer. 2006 Aug 1;6:202. doi: 10.1186/1471-2407-6-202. PMID 16882344
- [Background] Pignata S, Scambia G, Savarese A, Breda E, Sorio R, Pisano C, Lorusso D, Cognetti F, Vernaglia Lombardi A, Gebbia V, Scollo P, Morabito A, Signoriello G, Perrone F. Carboplatin and pegylated liposomal doxorubicin for advanced ovarian cancer: preliminary activity results of the MITO-2 phase III trial. Oncology. 2009;76(1):49-54. doi: 10.1159/000178760. Epub 2008 Nov 27. PMID 19039248
- [Result] Pignata S, Scambia G, Ferrandina G, Savarese A, Sorio R, Breda E, Gebbia V, Musso P, Frigerio L, Del Medico P, Lombardi AV, Febbraro A, Scollo P, Ferro A, Tamberi S, Brandes A, Ravaioli A, Valerio MR, Aitini E, Natale D, Scaltriti L, Greggi S, Pisano C, Lorusso D, Salutari V, Legge F, Di Maio M, Morabito A, Gallo C, Perrone F. Carboplatin plus paclitaxel versus carboplatin plus pegylated liposomal doxorubicin as first-line treatment for patients with ovarian cancer: the MITO-2 randomized phase III trial. J Clin Oncol. 2011 Sep 20;29(27):3628-35. doi: 10.1200/JCO.2010.33.8566. Epub 2011 Aug 15. PMID 21844495